CLINICAL TRIAL: NCT04720118
Title: Does Locus of Control Affect Satisfaction and Quality of Life During COVID - 19?
Brief Title: Parkinson's Disease and Experiences Throughout the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Towson University (Other)
Responsible Party: Principal Investigator, MacKenzie Forbes, Graduate Student, Towson University
Other Study IDs: 1352
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease; Covid19; Satisfaction, Patient; Quality of Life
MeSH Terms: conditions — Parkinson Disease; COVID-19; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study.

SUMMARY:
The purpose of this research study is to examine the relationship between personal characteristics and satisfaction with care in those diagnosed with Parkinson's disease during the COVID-19 pandemic. Participants will take 4 different surveys regarding their satisfaction with care throughout the duration of the COVID-19 pandemic. The surveys in total should not take more than 30 minutes to complete

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with Parkinson's Disease
* Must be able to complete the surveys without any help

Exclusion Criteria:

* Under the age of 18
* Not diagnosed with Parkinson's Disease
* Unable to complete the surveys without help

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is people, 18 years or older, who are diagnosed with Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Measure of the relationship between Locus of Control and Quality of Life | 1 year
  Participants will take the Multidimensional Health Locus of Control (MHLC) Scale. This will determine if the participant has more of an internal or external locus of control. Participants will also take the Quality of Life Scale- U.S Parkinson's Disease Questionnaire (PDQ-39) to determine the quality of life they have been experiencing throughout the COVID-19 pandemic. Based on the results of both surveys, the researchers will be able to determine if external locus of control or internal locus of control leads to a better quality of life in PD patients throughout the COVID-19 pandemic.
Measure of secondary control and satisfaction with care | 1 year
  Participants will take the Multidimensional Health Locus Control (MHLC) scale. This will determine what type of control is most present in the participant's life. Additionally, participant's will take the Short Form Patient Satisfaction Questionnaire (PSQ-18). This will determine how satisfied participants are with their healthcare providers throughout the COVID-19 pandemic. Based off of the responses to the surveys, the researcher will be able to determine whether a higher or lower secondary control yields a higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Towson University, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Qualtrics Link to the surveys for the study — http://towson.az1.qualtrics.com/jfe/form/SV_dp5NeNBH1K11Sp7